CLINICAL TRIAL: NCT07108608
Title: Treating OUD/PTSD in Residential Care: Written Exposure in Substance Treatment (WEST).
Brief Title: Adaptation of Written Exposure Therapy in Substance Treatment
Acronym: WEST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Potomac Health Foundations (Other)
Collaborators: University of Maryland, Baltimore County (Other)
Responsible Party: Principal Investigator, Rebecca Schacht, Affiliated Research Scientist, Potomac Health Foundations
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WEST 3.0
Record Dates: First submitted 2025-07-29; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Posttraumatic Stress Disorder; Substance Use Disorders
Keywords: Written Exposure Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Investigators are conducting an uncontrolled trial of approximately 20 subjects who will be assigned to adapted Written Exposure Therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAU + Adapted Written Exposure Therapy (WET) (Experimental): Participants in this condition receive everything included in TAU plus 5 individual sessions of WET delivered by a therapist. WET has been adapted for delivery in a residential SUD setting according to expert feedback. Sessions average less than 60 minutes and primarily involve writing about the traumatic experience that is guided by the therapist.
  Interventions: Behavioral: Written Exposure Therapy; Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Written Exposure Therapy — Written Exposure Therapy is a brief, evidenced based intervention for PTSD. WET is generally delivered individually across 5 sessions in which the therapist guides the patient through writing exercises. Across exposure sessions, participants experience habituation so that their symptoms decrease by the end of treatment. WET has an established evidence base in general outpatient psychotherapy for PTSD, but has not been adapted or tested in residential SUD treatment settings. Further, the investigators have adapted WET for this setting based on stakeholder and expert feedback.
Behavioral: Treatment as Usual — Treatment as Usual will include a variety of standard care services offered in short term residential treatment. For example, participants receiving TAU will participate in individual case management/general counseling sessions focused on substance use disorder and its consequences, group based psychoeducation sessions, group based counseling sessions (e.g., relapse prevention planning), individual services with a medical provider and pharmacotherapy (e.g., for withdrawal, relapse prevention, or co-occurring conditions)

SUMMARY:
The purpose of this pilot non-randomized, uncontrolled clinical trial is to test the feasibility and efficacy of written exposure therapy (WET) for posttraumatic stress disorder (PTSD) as adapted for use within the context of residential substance use disorder (SUD) treatment. All participants meet criteria for PTSD and are in a short term residential SUD treatment program (target residential treatment duration = 28 days) regardless of the research. The main question the study aims to answer is: 1) Is the delivery of adapted WET feasible and acceptable in short term residential SUD treatment for individuals with severe SUD?

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in residential SUD treatment at MTC
* Meet criteria for PTSD based on the Clinician-Administered PTSD Scale for DSM-5
* Be 18 years of age or older
* Have sufficient memory of the index trauma to write about it
* Be English speaking.

Exclusion Criteria:

* Inability to give informed consent for any reason (e.g., cognitive impairment)
* Presence of acute psychosis or suicidality that would interfere with study participation
* planning to leave residential treatment before WEST could realistically be completed as determined by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-25 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
PTSD symptom reduction | Pre-WEST intervention; post-WEST intervention (approximately 14 days after randomization, but will vary based on when participants complete the intervention); 4-weeks post enrollment; 8-weeks post enrollment; 12-weeks post enrollment.
  PTSD symptom reduction pre/post intervention by treatment arm as measured by the posttraumatic checklist for DSM-5 (PCL-5). The PCL-5 is a self-report questionnaire yielding scores ranging from 0-80 with higher scores indicating greater symptomology.

SECONDARY OUTCOMES:
Feasibility of WET delivered in residential SUD treatment context | Up to 4 weeks, or until the participant discharges from residential treatment (whichever comes first).
  Percentage of participants in the WET arm who were able to complete the treatment (5 sessions) prior to discharge
Acceptability of WET delivered in residential SUD treatment context | Collected post intervention window (approximately 3 weeks from enrollment)
  Treatment satisfaction scores among WET participants as measured by the 2-part credibility/expectancies questionnaire (CEQ). The CEQ utilizes two scoring systems that range from 1-9 or 0%-100%. with higher scores indicating greater acceptability.

CONTACTS AND LOCATIONS:
Locations (1):
- Maryland Treatment Centers, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD may be shared with other researchers through a de-identified, secure, electronic data transfer as allowed by the IRB and other regulatory authorities.
Time Frame: Interested individuals may inquire after data lock is achieved and the primary outcomes paper has been published from this dataset. Estimated time: 2026

REFERENCES:
- [Background] Schacht RL, Wenzel KR, Meyer LE, Mette M, Mallik-Kane K, Rabalais A, Berg SK, Fishman M. A pilot test of Written Exposure Therapy for PTSD in residential substance use treatment. Am J Addict. 2023 Sep;32(5):488-496. doi: 10.1111/ajad.13442. Epub 2023 Jun 17. PMID 37329251